CLINICAL TRIAL: NCT00620854
Title: A Dose Selection Study of Oral Recombinant Salmon Calcitonin (rsCT) in Normal, Healthy, Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UGL-OR0702; Bio-Kinetic No.: 96508
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — salmon calcitonin; Tablets; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- rsCTA (Experimental): Oral Tablet
  Interventions: Drug: Oral Tablet
- rsCTB (Experimental): Oral Tablet
  Interventions: Drug: Oral Tablet
- Fortical (Active Comparator): Nasal Spray
  Interventions: Drug: Recombinant Salmon Calcitonin (rsCT); Drug: Nasal Spray

INTERVENTIONS:
Drug: Recombinant Salmon Calcitonin (rsCT) — Single dose of a nasal spray or one of two doses of tablets, randomized to visits 2, 3, and 4.
  Other Names: Fortical® nasal spray
  Arms: Fortical
Drug: Oral Tablet — 0.15 mgs recombinant salmon calcitonin, single oral dose
  Arms: rsCTA
Drug: Oral Tablet — 0.2mgs recombinant salmon calcitonin, single oral tablet
  Arms: rsCTB
Drug: Nasal Spray — 200 IU recombinant salmon calcitonin, single intranasal spray
  Arms: Fortical

SUMMARY:
This study compares the performance of different doses of oral recombinant salmon calcitonin (rsCT).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, in good health (at least 5 years since last menses)
* Age ≥45 and ≤70
* Weight + or - 20% of the Metropolitan Life weight table
* Plasma C-terminal telopeptide of type I collagen (CTx-1) ≥ 0.25 ng/mL
* Total calcium (Ca++), phosphorus (P), and magnesium (Mg++) within normal range
* Willing and able to comply with all study requirements
* Willing and able to sign written informed consent
* Negative urine pregnancy test at screening
* Negative Screen for Hepatitis B and C, human immunodeficiency virus (HIV) and drugs of abuse

Exclusion Criteria:

* History of parathyroid, thyroid, pituitary or adrenal diseases
* History of musculoskeletal disease
* History of gastro-esophageal reflux disease (GERD) or other significant gastrointestinal disorders
* History of cancer within 5 years of enrollment other than basal cell carcinoma
* History of regular use of non-steroidal anti-inflammatory drugs (NSAID)
* History of surgery within 60 days of enrollment
* History of hypersensitivity or allergies (other than seasonal allergies) within 5 years of enrollment including known sensitivity to the active ingredients or the excipients in the study medications
* Use of concomitant medications other than acetaminophen within 7 days of enrollment or anticipated need to use such concomitant medications during the study
* Use of bisphosphonates within 6 months, selective selective estrogen receptor modulators (SERMS), estrogen or estrogen-like drugs 2 months, or calcitonin 1 month
* Presence of any clinically significant illness
* Unwilling or unable to comply with all study requirements
* Unwilling or unable to sign written, informed consent
* History of drug or alcohol abuse
* Participation in any clinical study of an investigational drug within 60 days of enrollment
* Plasma CTx-1 less than 0.25 ng/mL

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Legg, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the study site data base during January 2008.
Groups:
- rsCTA Then rsCTB Then Fortical; rsCTA Then Fortical Then rsCTB; rsCTB Then rsCTA Then Fortical; rsCTB Then Fortical Then rsCTA; Fortical Then rsCTA Then rsCTB; Fortical Then rsCTB Then rsCTA: single dose rsCTA tablets (150 micrograms), single dose rsCTB tablets (200 micrograms), Fortical nasal spray (200 IU)
Period: Period 1
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Period: Period 2
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Started | 4 | 4 | 3 | 3 | 4 | 4
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Started | 4 | 4 | 3 | 3 | 4 | 4
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Started | 4 | 4 | 3 | 3 | 4 | 4
Completed | 4 | 4 | 3 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 3 | 4 | 4 | 4 | 21
  >=65 years | 0 | 2 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 4 | 4 | 24
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Plasma C-terminal Telopeptide of Type I Collagen (CTx-1)(% Change From Baseline)
Description: This study compared the exposure to recombinant salmon calcitonin (rsCT), as measured by a decrease in plasma C-terminal telopeptide of type I collagen (CTx-1), of single doses of rsCT tablets containing 150 µg and 200 µg rsCT, respectively, with Fortical® nasal spray.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, and 24 hours (Fortical): 0, 2, 3, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 10, 12, 24 hours rsCTA and rsCTB
Population: Per protocol, only subjects who completed all 3 treatments were analyzed.
Measure: Mean (Standard Error); unit: % Change in Baseline CTx-1
Groups:
- rsCT A: Oral rsCT (150 micrograms)
- rsCTB: Oral rsCT (200 micrograms)
- Fortical®: Fortical nasal spray (200 IU)
Arm/Group | rsCT A | rsCTB | Fortical®
Number analyzed (Participants) | 22 | 22 | 22
% Change in Baseline CTx-1 | -74.17 (2.44) | -71.99 (2.88) | -68.40 (2.80)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at each study visit. The three study periods occurred at weekly intervals, so the AE data were collected over a period of 3 weeks.
Arm/Group | rsCTA Then rsCTB Then Fortical | rsCTA Then Fortical Then rsCTB | rsCTB Then rsCTA Then Fortical | rsCTB Then Fortical Then rsCTA | Fortical Then rsCTA Then rsCTB | Fortical Then rsCTB Then rsCTA
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 1/4 | 1/4 | 3/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rsCTA Then rsCTB Then Fortical (N=4) | rsCTA Then Fortical Then rsCTB (N=4) | rsCTB Then rsCTA Then Fortical (N=4) | rsCTB Then Fortical Then rsCTA (N=4) | Fortical Then rsCTA Then rsCTB (N=4) | Fortical Then rsCTB Then rsCTA (N=4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction is that the Principal Investigator (PI) cannot without the sponsor's prior written consent, transmit, publish, or otherwise disclose to any person or entity either clinical trial results information.